CLINICAL TRIAL: NCT00014976
Title: Spasticity: Physiologic Studies
Brief Title: Physiologic Studies of Spasticity
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010148; 01-N-0148
Record Dates: First submitted 2001-04-17; First posted 2001-04-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-11-01

CONDITIONS: Muscle Spasticity; Healthy
Keywords: Pyramidal Tract; Primary Lateral Sclerosis; Spastic Paraparesis; EMG; Magnetic Stimulation; Muscle Spasticity; Healthy Volunteer
MeSH Terms: conditions — Muscle Spasticity; Motor Neuron Disease; Paraparesis, Spastic

SUMMARY:
This study will provide information about changes that occur in the motor neurons of the spinal cord (the nerve cells that control the muscles) when the motor cortex (the region of the brain that controls movement) is unable to send messages to the spinal cord and muscles in the normal way. This information will help elucidate how the nervous system adapts after injury or disease of the motor cortex.

Healthy adult volunteers and adults with a spasticity disorder and moderate weakness may be eligible for this study. Patients will be screened with a medical history, physical examination and diagnostic studies as needed. Healthy volunteers will have a neurological examination. Muscle weakness and spasticity will be evaluated in both groups of subjects.

All participants will have electromyography (measurement of electrical activity in muscles) during nerve stimulation and transcranial magnetic stimulation, described below. (Some patients, such as those with a pacemaker or implanted medication pumps, metal objects in the eye, history of epilepsy and others, will not have magnetic stimulation.)

Electromyography - The electrical activity of muscles will be measured either by 1) using metal electrodes taped to the skin overlying a muscle, or 2) using thin wires inserted into the muscle through a needle.

Nerve stimulation - The nerves will be stimulated by applying a small electrical pulse through metal disks on the skin of the arm or leg.

Transcranial magnetic stimulation - A brief electrical current is passed through a wire coil placed on the scalp. This creates a magnetic pulse, which stimulates the brain. During the test, the participant may be asked to tense certain muscles slightly or perform other simple actions.

Nerve block - Some patients will have a nerve block of one of the nerves in the arm. For this procedure, a local anesthetic is injected under the skin to produce numbness and weakness in some arm muscles.

DETAILED DESCRIPTION:
Objective: The purpose of this protocol is to characterize abnormalities in motoneuron recruitment in adult patients with corticospinal tract dysfunction using electrophysiologic measures. We wish to determine whether the intrinsic spinal mechanisms for recruitment are abnormal or whether only inputs to motoneurons are changed. This information is pertinent for assessing ways that can ultimately be used to enhance strength in patients with corticospinal tract dysfunction using the existing spinal circuitry.

Study Design: Comparison of physiological observations in patients and age - matched control subjects.

Study Population: Adults with spastic paresis aged 21-80 and healthy volunteers.

Outcome Parameters: Measures of motor unit firing in response to peripheral nerve stimulation and transcranial magnetic stimulation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Adult patients with selective corticospinal tract dysfunction

Minimum age 21 years; maximum age 80 years

Moderate severity of weakness (greater than or equal to MRC Grade 4)

Adult normal volunteers

EXCLUSION CRITERIA:

Severe weakness with inability to maintain voluntary contractions

Significant sensory impairment

For TMS studies only: pregnancy, implanted devices such as pacemakers, medication pumps or defibrillators, metal in the cranium except the mouth, intracardiac lines, history of seizures

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2001-04-13; Study Completion 2010-11-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gemperline JJ, Allen S, Walk D, Rymer WZ. Characteristics of motor unit discharge in subjects with hemiparesis. Muscle Nerve. 1995 Oct;18(10):1101-14. doi: 10.1002/mus.880181006. PMID 7659104
- [Background] Rosenfalck A, Andreassen S. Impaired regulation of force and firing pattern of single motor units in patients with spasticity. J Neurol Neurosurg Psychiatry. 1980 Oct;43(10):907-16. doi: 10.1136/jnnp.43.10.907. PMID 7441270
- [Background] Frascarelli M, Mastrogregori L, Conforti L. Initial motor unit recruitment in patients with spastic hemiplegia. Electromyogr Clin Neurophysiol. 1998 Jul-Aug;38(5):267-71. PMID 9741003